CLINICAL TRIAL: NCT00402246
Title: CONNECT Study - Clinical Evaluation Of Remote NotificatioN to rEduCe Time to Clinical Decision
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Symbios Clinical (Other)
Responsible Party: CONNECT Trial Leader, Medtronic, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 605
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2011-02-16 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Arrhythmia; Tachycardia; Atrial Fibrillation; Ventricular Fibrillation
Keywords: Randomized Controlled Trials; Defibrillators; Remote Consultation
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia; Atrial Fibrillation; Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote Arm (Experimental): Remote Management
  Interventions: Other: Remote Management
- In-office Arm (Active Comparator): In-Office Care
  Interventions: Other: In-Office Care

INTERVENTIONS:
Other: Remote Management — The Remote Management method of treating patients consists of 3 components:
  CareAlerts: Device alerts that are triggered by either device integrity issues or arrhythmic issues with the patient (e.g. multiple shocks delivered for a ventricular arrhythmia, more than 12 hours of atrial arrhythmias occurring in a day)
  Conexus: the device feature which allows the device to wirelessly transmit information (possibly triggered by a CareAlert) to a patient monitor that is hooked up a patient's phone line
  CareLink: the Medtronic system which allows device data to be transmitted from a patient's monitor through the phone line to ultimately be displayed on a secure website for viewing by the patient's physician.
  The combination of these 3 components allow the patient's device to transmit information relating to either a device issue or patient issue to be viewed by a clinician without the patient having to take direct action.
  Arms: Remote Arm
Other: In-Office Care — Routine in-office care
  Arms: In-office Arm

SUMMARY:
The purpose of this study is to determine whether the ability of clinicians to receive and review information from patients implanted with a heart device over the internet (remote care) is comparable to patients who are seen in-office for routine visits to check the status of their device.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be implanted with a Medtronic Conexus-enabled Cardiac Resynchronization Therapy Defibrillator (CRT-D) or Implantable Cardioverter-Defibrillator (DR-ICD) device.

Exclusion Criteria:

* Patient has permanent rapid beats in the upper chamber of the heart (Atrial Fibrillation) - (constant atrial fibrillation in which pharmacological therapy or cardioversion failed or not attempted).
* Patient plans to be on chronic warfarin therapy post-implant and is no longer receiving therapies to attempt to control the rhythm of the beats in their atrium.
* Patient has a previous ICD, CRT-D, Implantable Pulse Generator (IPG) or Cardiac Resynchronization Therapy Pacemaker (CRT-P).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2009 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Crossley, M.D., Principal Investigator — Mid-State Cardiology
Locations (127):
- United States (127):
  - Mobile, Alabama
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Fort Smith, Arkansas
  - Little Rock, Arkansas
  - East Palo Alto, California
  - Inglewood, California
  - Los Angeles, California
  - Napa, California
  - Rancho Mirage, California
  - San Bernardino, California
  - San Diego, California
  - Santa Rosa, California
  - Colorado Springs, Colorado
  - Bridgeport, Connecticut
  - Washington D.C., District of Columbia
  - Brooksville, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Lakeland, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Safety Harbor, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Gainesville, Georgia
  - Aurora, Illinois
  - Chicago, Illinois
  - Kankakee, Illinois
  - Moline, Illinois
  - Rockford, Illinois
  - Springfield, Illinois
  - Bloomington, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Ames, Iowa
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Ashland, Kentucky
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Covington, Louisiana
  - Baltimore, Maryland
  - Glen Burnie, Maryland
  - Lanham, Maryland
  - Randallstown, Maryland
  - Salisbury, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Chelmsford, Massachusetts
  - Ann Arbor, Michigan
  - Grand Blanc, Michigan
  - Petoskey, Michigan
  - Saginaw, Michigan
  - Saint Joseph, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Hattiesburg, Mississippi
  - Columbia, Missouri
  - Mexico, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Kearney, Nebraska
  - Omaha, Nebraska
  - Manchester, New Hampshire
  - Cherry Hill, New Jersey
  - Newark, New Jersey
  - Ridgewood, New Jersey
  - Wayne, New Jersey
  - West Orange, New Jersey
  - Flushing, New York
  - Mineola, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Williamsville, New York
  - Gastonia, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Fairview Park, Ohio
  - Kettering, Ohio
  - Mayfield Heights, Ohio
  - Whitehall, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Abington, Pennsylvania
  - Doylestown, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Langhorne, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wormleysburg, Pennsylvania
  - Wyomissing, Pennsylvania
  - York, Pennsylvania
  - Columbia, South Carolina
  - Florence, South Carolina
  - Greenwood, South Carolina
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Fairfax, Virginia
  - Fredericksburg, Virginia
  - Lynchburg, Virginia
  - Portsmouth, Virginia
  - Morgantown, West Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Crossley GH, Boyle A, Vitense H, Chang Y, Mead RH; CONNECT Investigators. The CONNECT (Clinical Evaluation of Remote Notification to Reduce Time to Clinical Decision) trial: the value of wireless remote monitoring with automatic clinician alerts. J Am Coll Cardiol. 2011 Mar 8;57(10):1181-9. doi: 10.1016/j.jacc.2010.12.012. Epub 2011 Jan 20. PMID 21255955
- [Derived] Crossley G, Boyle A, Vitense H, Sherfesee L, Mead RH. Trial design of the clinical evaluation of remote notification to reduce time to clinical decision: the Clinical evaluation Of remote NotificatioN to rEduCe Time to clinical decision (CONNECT) study. Am Heart J. 2008 Nov;156(5):840-6. doi: 10.1016/j.ahj.2008.06.028. Epub 2008 Sep 11. PMID 19061696

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first enrollment occurred 29 November 2006. A total of 1997 subjects were enrolled (i.e. consented, implanted, and randomized) in the study from a total of 136 activated clinical study centers.
Pre-assignment Details: There were an additional 12 patients (for a total of 2009 patients) consented for whom proper permission to use their data could not be obtained. Any data obtained for these patients was excluded from all reporting.
Groups:
- Remote Arm: Wireless remote monitoring, consisting of 3 components:
  CareAlerts: Device alerts that are triggered by either device integrity issues or arrhythmic issues with the patient (e.g. multiple shocks delivered for a ventricular arrhythmia, more than 12 hours of atrial arrhythmias occurring in a day)
  Conexus: the device feature which allows the device to wirelessly transmit information (possibly triggered by a CareAlert) to a patient monitor that is hooked up a patient's phone line
  CareLink: the Medtronic system which allows device data to be transmitted from a patient's monitor through the phone line to ultimately be displayed on a secure website for viewing by the patient's physician.
  The combination of these 3 components allow the patient's device to transmit information relating to either a device issue or patient issue to be viewed by a clinician without the patient having to take direct action.
- In-Office Arm: In-office care, consisting of standard follow-up procedures for a device patient such as review of the patient's device data during a patient's scheduled in-office visit
Period: Overall Study
Arm/Group | Remote Arm | In-Office Arm
Started | 1014 | 983
Completed | 794 | 749
Not Completed | 220 | 234
Not completed — Death | 62 | 58
Not completed — Lost to Follow-up | 20 | 28
Not completed — Withdrawal by Subject | 72 | 87
Not completed — Physician Decision | 24 | 26
Not completed — Protocol Violation | 25 | 24
Not completed — Missed Final Visit | 1 | 2
Not completed — Insurance Issues | 2 | 1
Not completed — Heart Transplant | 0 | 1
Not completed — Patient's device explanted | 6 | 2
Not completed — Center Closure | 5 | 3
Not completed — Deterioriating Condition | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Arm | In-Office Arm | Total
Number analyzed (Participants) | 1014 | 983 | 1997
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 453 | 442 | 895
  >=65 years | 561 | 540 | 1101
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (12.4) | 64.9 (11.9) | 65.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299 | 278 | 577
  Male | 715 | 705 | 1420
Region of Enrollment [Number; unit: participants]
  United States | 1014 | 983 | 1997

OUTCOME MEASURES:

1. Primary Outcome: Time Per Patient From a Clinical Event to a Clinical Decision in Response to Arrhythmias, Cardiovascular (CV) Disease Progression, and Device Issues
Description: Days from device detection of a clinical event to a decision being made in response to the event, as reported by the clinician or as evidenced by device data obtained at interrogation. A clinical event could be any of the following that satisfied pre-specified thresholds: arrhythmias (e.g. at least 12 hours of atrial tachycard/atrial fibrillation in a day), cardiovascular disease progression (e.g. multiple device shocks delivered to terminate a single episode), or device issues (e.g. low battery).
Time Frame: Enrollment to last visit (up to 15 month post-implant)
Population: All enrolled subjects who experienced at least one event and satisfied the inclusion/exclusion criteria were included in the analysis. An intention to treat analysis was performed for this objective.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 172 | 145
days | 4.6 [1.0 to 13.3] | 22.0 [7.0 to 44.2]
Statistical Analysis 1: Comparison: Remote Arm vs In-Office Arm; The null hypothesis is that the time from a clinical event to a clinical decision for patients followed through the remote management system is greater than and equal to that of patients receiving only in-office care; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — The a priori threshold for significance was an alpha level of 0.05; Median Difference (Final Values) = 17.4

2. Secondary Outcome: Health Care Utilization (HCU)
Description: Count of HCU visits for each HCU type (cardiovascular (CV) hospitalizations, cardiovascular (CV) emergency department (ED), and cardiovascular (CV) unscheduled clinic office/urgent care visits)
Time Frame: Enrollment to last visit (up to 15 month post-implant)
Population: 9 remote arm patients and 8 in-office arm patients did not meet the inclusion/exclusion criteria. The remaining 1005 remote arm patients and 975 in-office arm patients were included in the analysis. An intention to treat analysis was performed for this objective.
Measure: Number; unit: Visits
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 1005 | 975
Visits
  CV hospitalizations | 567 | 508
  Emergency department (ED) | 270 | 223
  CV unscheduled clinic office/urgent care visits | 2545 | 2114
Statistical Analysis 1: Comparison: Remote Arm vs In-Office Arm; An Andersen-Gill proportional hazards regression model was fit to test the hypothesis that the CV hospitalization hazard rates for patients in the remote arm is equal to that of similar patients in the in-office arm; Test type: Superiority or Other; p = 0.524, Andersen-Gill model — Model was fit with device group (CRT-D vs. DR-ICD) as a stratifying variable; An Andersen-Gill model was utilized to account for multiple hospitalization events per subject; Hazard Ratio (HR) = 1.06, 95% CI 1-sided [upper limit 1.21]
Statistical Analysis 2: Comparison: Remote Arm vs In-Office Arm; An Andersen-Gill proportional hazards regression model was fit to test the hypothesis that the ED hazard rates for patients in the remote arm is equal to that of similar patients in the in-office arm; Test type: Superiority or Other; p = 0.325, Andersen-Gill model — Model was fit with device group (CRT-D vs. DR-ICD) as a stratifying variable; An Andersen-Gill model was utilized to account for multiple ED visits per subject; Hazard Ratio (HR) = 1.14, 95% CI 1-sided [upper limit 1.43]
Statistical Analysis 3: Comparison: Remote Arm vs In-Office Arm; An Andersen-Gill proportional hazards regression model was fit to test the hypothesis that the hazard rates of the CV unscheduled clinic or urgent care visits for patients in the remote arm is equal to that of similar patients in the in-office arm; Test type: Superiority or Other; p = 0.099, Andersen-Gill model — Model was fit with device group (CRT-D vs. DR-ICD) as a stratifying variable; An Andersen-Gill model was utilized to account for multiple unscheduled clinic visits per subject; Hazard Ratio (HR) = 1.14, 95% CI 1-sided [upper limit 1.31]

3. Secondary Outcome: Health Care Utilization: TEEs
Description: Count of Transesophageal echocardiograms (TEEs) performed
Time Frame: Enrollment to last visit (up to 15 months post-implant)
Population: as for outcome 2
Measure: Number; unit: Procedures
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 1005 | 975
Procedures | 26 | 17
Statistical Analysis 1: Comparison: Remote Arm vs In-Office Arm; An Andersen-Gill proportional hazards regression model was fit to test the hypothesis that the hazard rate of transesophageal echocardiography (TEE) taken for patients in the remote arm is equal to that of similar patients in the in-office arm; Test type: Superiority or Other; p = 0.29, Andersen-Gill model — Model was fit with device group (CRT-D vs. DR-ICD) as a stratifying variable; Hazard Ratio (HR) = 1.45, 95% CI 1-sided [upper limit 2.56]

4. Secondary Outcome: Actions Taken for HCU Visits
Description: Count of HCU visits that involved specific actions taken
Time Frame: Enrollment to last visit (up to 15 month post-implant)
Measure: Number; unit: Visits
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 1005 | 975
Visits
  Total # of HCU visits | 3869 | 2895
  Total # of HCU visits with no Action Taken | 687 | 513
  Total # of HCU visits with TEE | 26 | 17
  Total # of HCU visits with Echo | 221 | 218
  Total # of HCU visits with EKG | 670 | 514
  Total # of HCU visits with device interrogation | 903 | 531
  #of HCU visits with oral CV medication change | 771 | 710
  # of HCU visits with IV CV medication administered | 225 | 194
  Total # of HCU visits with device reprogramming | 429 | 170
  #of HCU visits with surgical/invasive procedure | 60 | 54
  Total # of HCU visits with system modification | 32 | 56
  Total # of HCU visits with diagnostic test ordered | 298 | 260
  Total # of HCU visits with calling subject | 137 | 3
  Total # of HCU visits with bringing into clinic | 143 | 27
  # of HCU visits with referring to another clinic | 85 | 52
  Total # of HCU visits with admission to hospital | 197 | 150
  # of HCU visits with waiting till next clinic appt | 41 | 29
  Total # of HCU visits with sending to ED | 12 | 5
  Total # of HCU visits with blood test(s) | 1089 | 1004
  Total # of HCU visits with chest x-ray | 380 | 328
  Total # of HCU visits with exercise testing | 36 | 23
  Total # of HCU visits with EP study | 16 | 11
  Total # of HCU visits with cardioversion | 37 | 22
  Total # of HCU visits with other imaging | 76 | 76
  Total # of HCU visits with wound check | 130 | 111
  Total # of HCU visits - other action taken | 396 | 285
  #of HCU visits with defibrillation threshold test | 116 | 68
  #of HCU visits with pacing threshold testing | 341 | 213
  #of HCU visits with other device testing | 130 | 89

5. Secondary Outcome: Clinically Meaningful Alerts
Description: Count of clinically meaningful alerts as classified by the clinician
Time Frame: Enrollment to last visit (up to 15 month post-implant)
Population: All enrolled remote subjects who experienced at least one alert were included in the analysis. Alerts that were not classified by the clinician as clinically meaningful or not were excluded from the analysis.
Measure: Number; unit: Alerts
Units Other Than Participants: Events
Arm/Group | Remote Arm
Number analyzed (Participants) | 170
Number analyzed (Events) | 379
Alerts | 238

6. Secondary Outcome: Symptomatic AT/AF Alerts
Description: AT/AF represents atrial tachycardia or atrial fibrillation which are arrhythmias involving rapid beating of the atrial chambers of the heart. The devices in this study store how many hours each day that a patient experiences AT/AF. The patient may not be aware they are experiencing these atrial arrhythmias, but if the AT/AF is accompanied by symptoms, the AT/AF is said to be symptomatic AT/AF. Devices in this study have an alert that fires if the patient experiences at least a programmed amount of AT/AF in a day. Measure is count of symptomatic AT/AF alerts as classified by the clinician
Time Frame: Enrollment to last visit (up to 15 month post-implant)
Population: All enrolled remote patients who experienced at least one AT/AF alert were included in the analysis. AT/AF alerts there were not classified by the clinician as symptomatic or asymptomatic were excluded from the analysis.
Measure: Number; unit: Alerts
Units Other Than Participants: Events
Arm/Group | Remote Arm
Number analyzed (Participants) | 107
Number analyzed (Events) | 255
Alerts | 73
Statistical Analysis 1: Comparison: Remote Arm; Test type: Superiority or Other; Regression, Logistic; A GEE model was utilized to account for multiple events within same patient in estimating the probability of an AT/AF alert event being symptomatic; probability = 0.23

7. Secondary Outcome: AT/AF Alert Treatment
Description: Count of the treatment (i.e. hospitalization, ED visit, unscheduled clinic office/urgent care visits) in response to the AT/AF alerts
Time Frame: Enrollment to last visit (up to 15 month post-implant)
Population: All enrolled remote patients who had at least one AT/AF alert were included in the analysis.
Measure: Number; unit: Alerts
Units Other Than Participants: Events
Arm/Group | Remote Arm
Number analyzed (Participants) | 112
Number analyzed (Events) | 287
Alerts
  No Treatment | 159
  ED | 2
  Hospitalization | 23
  Unscheduled Clinic Office/Urgent Care Visits | 89
  Other Treatment | 30

8. Secondary Outcome: Time Per Patient From a Clinical Event Onset to a Clinical Decision for Symptom-driven Device Interrogations
Description: Days from a symptom-driven device interrogation event onset to a clinical decision being made in response to the event as reported by the clinician. An event is defined as a subject complaint received by the managing clinician in which the clinician determines that he/she must interrogate the subject's device to properly treat the subject.
Time Frame: Enrollment to last visit (up to 15 month post-implant)
Population: All enrolled subjects who experienced at least one event and satisfied the inclusion/exclusion criteria were included in the analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 208 | 154
Days | 0.8 (4.9) | 0.7 (3.3)
Statistical Analysis 1: Comparison: Remote Arm vs In-Office Arm; The null hypothesis is that the time from event onset to clinical decision for symptom-driven device interrogations for patients followed through the remote management system is greater than and equal to that of patients receiving only in-office care; Test type: Superiority or Other; p = 0.779, t-test, 2 sided — The a priori threshold for significance was an alpha level of 0.05; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.8 to 1.0], Standard Deviation 4.3

9. Secondary Outcome: Time Per Patient From a Clinical Event Onset to a Clinical Decision for Both Device Events and Symptom-driven Device Interrogations
Description: Days from device detection of a clinical event or a symptom-driven device interrogation event onset to a clinical decision, as reported by the clinician or as evidenced by device data obtained at interrogation. A clinical event is an event as defined in the primary objective. A symptom-driven device interrogation event is defined as a subject complaint received by the managing clinician in which the clinician determines that he/she must interrogate the subject's device to properly treat the subject.
Time Frame: From event onset to clinical decision
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 324 | 265
Days | 6.7 (13.3) | 16.7 (24.4)
Statistical Analysis 1: Comparison: Remote Arm; The null hypothesis is the time from event onset to clinical decision for both device events and symptom-driven device interrogations for patients followed through the remote management system is greater than and equal to that of patients receiving only in-office care; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The a priori threshold for significance was an alpha level of 0.05; Mean Difference (Final Values) = -10.0, 95% CI 2-sided [-13.1 to -6.9], Standard Deviation 19.1

10. Other Pre Specified Outcome: Length of Hospital Stay (LOS)
Description: LOS per cardiovascular hospitalization
Time Frame: Enrollment to last visit (up to 15 month post-implant)
Population: All enrolled subjects who satisfied the inclusion/exclusion criteria and had at least one cardiovascular hospitalization were included in the analysis.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 336 | 333
Days | 3.3 (0.15) | 4.0 (0.18)
Statistical Analysis 1: Comparison: Remote Arm vs In-Office Arm; The null hypothesis was that the mean LOS per hospitalization visit for patients in the remote arm was equal to that for similar patients in the in-office arm; Test type: Superiority or Other; p = 0.002, negative binomial model — The a priori threshold for statistical significance was 0.05. The threshold was met, and the null hypothesis was rejected; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.7 to 0.9]

11. Secondary Outcome: CareLink Transmission Compliance
Description: The CareLink Transmission Compliance Rate for a particular visit (e.g. 3 month visit) is the proportion (ranging from 0 to 1) of subjects with device interrogation data remotely transmitted via the CareLink system on the date it was scheduled to be sent for that visit. The proportion is a fraction in which the denominator is the number of subjects in the Remote Arm who were not exited from the trial prior to the visit of interest, and the numberator is the number of Remote Arm subjects who successfully transmitted device data via the CareLink system on the date it was scheduled to be sent.
Time Frame: 3, 6, 9, 12 months visits
Population: 9 of 1014 remote arm subjects did not meet the inclusion/exclusion criteria and were excluded from the analysis. The remaining 1005 remote arm subjects were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Remote Arm
Number analyzed (Participants) | 1005
Proportion of subjects
  3 Month CareLink Transmission Compliance Rate | 0.761 [0.737 to 1.00]
  6 Month CareLink Transmission Compliance Rate | 0.815 [0.793 to 1.00]
  9 Month CareLink Transmission Compliance Rate | 0.815 [0.792 to 1.00]
  12 Month CareLink Transmission Compliance Rate | 0.814 [0.790 to 1.00]
Statistical Analysis 1: Comparison: Remote Arm; 3-month compliance rate; Test type: Superiority or Other; Binomial Exact Test; compliance rate = 0.761, 95% CI 1-sided [lower limit 0.737]
Statistical Analysis 2: Comparison: Remote Arm; 6-month compliance rate; Test type: Superiority or Other; Binomial Exact Test; compliance rate = 0.815, 95% CI 1-sided [lower limit 0.793]
Statistical Analysis 3: Comparison: Remote Arm; 9-month compliance rate; Test type: Superiority or Other; Binomial Exact Test; compliance rate = 0.815, 95% CI 1-sided [lower limit 0.792]
Statistical Analysis 4: Comparison: Remote Arm; 12-month compliance rate; Test type: Superiority or Other; Binomial Exact Test; compliance rate = 0.814, 95% CI 1-sided [lower limit 0.79]

12. Secondary Outcome: Variability in Left Ventricular (LV) Threshold as Measured by Left Ventricular Capture Management (LVCM)
Description: LV Capture Threshold is the required energy(volts) necessary to cause the left ventricule to contract. It is important that a device which paces the left ventricule be set to a threshold such that current conducted through the left ventricular lead will induce contraction in the left ventricle. However, these thresholds may vary over time.
  The standard deviation and range (maximum LVCM threshold - minimum LVCM threshold) of the most recent 14 days of LVCM results prior to each follow-up visit were determined for each subject and used to assess within-patient variability in LV thresholds.
Time Frame: 1, 3, 6, 9, 12, and 15 months visits
Population: All enrolled subjects who were implanted with a Concerto CRT-D (Cardiac Resynchronization Therapy with Defibrillation)device, met inclusion/exclusion criteria, and had daily LVCM measurement for at least one of the 6 scheduled visits/transmissions were included in the analysis.
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Patients With a Study CRT-D Device: Patients in either the Remote Arm or the In-office Arm who were implanted with a study CRT-D Device, as these are the only devices that have Left Ventricular leads
Arm/Group | Patients With a Study CRT-D Device
Number analyzed (Participants) | 604
Volts
  1 month standard deviation | 0.181 (0.202)
  3 month standard deviation | 0.117 (0.142)
  6 month standard deviation | 0.118 (0.138)
  9 month standard deviation | 0.121 (0.154)
  12 month standard deviation | 0.132 (0.142)
  15 month standard deviation | 0.135 (0.149)
  1 month range | 0.500 (0.606)
  3 month range | 0.324 (0.418)
  6 month range | 0.326 (0.419)
  9 month range | 0.345 (0.476)
  12 month range | 0.374 (0.428)
  15 month range | 0.381 (0.459)

13. Secondary Outcome: State-Anxiety Scale
Description: The State-Anxiety scales for each subject were obtained at multiple time points. The State-Anxiety scale was derived by summing the 20 scores in the State section of the State-Trait Anxiety Inventory (STAI) questionnaire. The State-Anxiety scales can vary from a minimum of 20 (best possible) to a maximum of 80 (worst possible).
Time Frame: 1, 3, 6, 9, 12, and 15 month visit
Population: All enrolled subjects who completed the STAI questionnaire for all scheduled follow-up visits/transmissions that occurred within specified visit windows and satisfied the inclusion/exclusion criteria were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 484 | 419
Scores on a scale
  1 month | 31.0 (10.9) | 32.1 (12.0)
  3 month | 30.3 (10.6) | 31.6 (11.8)
  6 month | 30.0 (11.1) | 30.7 (11.0)
  9 month | 30.5 (11.5) | 30.6 (11.2)
  12 month | 30.2 (11.7) | 31.2 (12.0)
  15 month | 31.0 (12.4) | 32.7 (12.8)
Statistical Analysis 1: Comparison: Remote Arm vs In-Office Arm; A mixed model was fit to test whether patients followed through the remote management system will experience less anxiety than patients followed through in-office care; Test type: Superiority or Other; p = 0.217, Mixed Models Analysis — The a prior threshold for statistical significance was 0.05; Model was fit with randomization arm, device group (CRT-D vs. DR-ICD), and follow-up visit as fixed effects, and subject as a random effect

14. Secondary Outcome: Trait-Anxiety Scale
Description: The Trait-Anxiety scales for each subject were obtained at multiple time points. The Trait-Anxiety scale was derived by summing the 20 scores in the Trait section of the STAI questionnaire. The Trait-Anxiety scales can vary from a minimum of 20 (best possible) to a maximum of 80 (worst possible).
Time Frame: 1, 3, 6, 9, 12, and 15 months visits
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Remote Arm | In-Office Arm
Number analyzed (Participants) | 459 | 393
Scores on a scale
  1 month | 31.2 (10.5) | 32.1 (11.4)
  3 month | 29.8 (9.6) | 31.3 (11.3)
  6 month | 29.6 (10.3) | 30.8 (10.7)
  9 month | 29.7 (10.6) | 30.6 (10.9)
  12 month | 29.6 (10.7) | 30.5 (11.5)
  15 month | 30.7 (11.1) | 30.8 (11.6)
Statistical Analysis 1: Comparison: Remote Arm vs In-Office Arm; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.154, Mixed Models Analysis — The a priori threshold for statistical significance for was 0.05; [statistical method as in outcome 13, analysis 1]

15. Secondary Outcome: Clinic Personnel Satisfaction With Wireless Telemetry (Telemetry + Leadless ECG).
Description: Following the completion of enrollment in the study, participating clinicians were asked to complete a survey assessing their overall satisfaction with the wireless telemetry feature. Clinicians' rating (1=strongly disagree, 5=strongly agree) of the overall satisfaction with the wireless telemetry feature of the device
Time Frame: After study enrollment has been completed; on average 15.8 months after the center had enrolled its first subject
Population: All surveys in which clinician completed at least a subset of the questions were included.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Clinicians: Clinicians who responded to the survey
Arm/Group | Clinicians
Number analyzed (Participants) | 212
Units on a scale
  Satisfaction with the Full-Wireless follow-up | 4.3 (0.8)
  Prefer to perform wireless follow-up | 4.0 (1.0)
  Prefer to use leadless ECG during follow-up | 3.8 (1.0)
  Pts were more comfortable with wireless follow-up | 4.2 (1.0)
  Treated pts sooner due to wireless CareAlerts | 4.0 (0.9)
  Provided better pt care due to wireless CareAlerts | 3.9 (0.9)

16. Secondary Outcome: In-office Follow-up Burden: Distance Traveled
Description: Subjects' responses to the survey. Subjects were asked to provide the distance (in miles) from their home to the clinic/hospital.
Time Frame: 1 month visit
Population: All enrolled subjects who completed some portion of the caregiver burden survey and satisfied the inclusion/exclusion criteria were included.
Measure: Mean (Standard Deviation); unit: Miles
Groups:
- Enrolled Subjects: All enrolled subjects who completed some portion of the caregiver burden survey at 1 month visit
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 1854
Miles | 49.2 (63.4)

17. Secondary Outcome: In-office Follow-up Burden: Patient Expenses
Description: On a survey at the one month visit, the patient estimated their expenses in traveling to that visit.
Time Frame: 1 month
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 1854
Dollars | 15.0 (21.0)

18. Secondary Outcome: In-office Follow-up Burden: Hours Absent From Work Due to Visit
Description: Subjects were asked at their one month visit to indicate on a survey how many hours of work they were missing to attend that visit.
Time Frame: 1 month
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 1854
Hours | 4.4 (3.5)

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected in the CONNECT Study.
Description: Products used in the study were market approved and used within labeling indications. Centers were instructed to report Unanticipated Adverse Device Events(UADE) in the manner required for any commercially available device: through the Medical Device Reporting(MDR) processes and in accordance with any reporting requirements required by their IRB.
Groups:
- Enrolled Subjects: All enrolled subjects in the study
Arm/Group | Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigational Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication.